CLINICAL TRIAL: NCT02025075
Title: A Prospective, Double-blind, Randomized, Crossover Design Study to Compare the Hemodynamic and Respiratory Variations During Laparoscopic Surgery in Patients With and Without Deep Neuromuscular Blockade.
Brief Title: Hemodynamic and Respiratory Variations During Laparoscopic Surgery With and Without Deep Neuromuscular Blockade.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marcos Vidal Melo, Associate Professor of Anesthesia, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Merck-50706
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Intraoperative Complications; Postoperative Complications; Laparoscopy; Surgical Complications From General Anesthesia; Ventilator-Induced Lung Injury
Keywords: Tomography; Oximetry; Echocardiography
MeSH Terms: conditions — Intraoperative Complications; Postoperative Complications; Ventilator-Induced Lung Injury | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Neuromuscular Block (NMB) (Experimental): Muscle paralysis with rocuronium 0.6 - 1.2 mg/kg with the dose adjusted to achieve 1-2 post-tetanic counts (neuromuscular function monitor).
  Interventions: Drug: Rocuronium
- Moderate Neuromuscular block (NMB) (Active Comparator): Muscle paralysis with rocuronium 0.6 - 1.2 mg/kg with the dose adjusted to achieve 1-2 twitches in the train-on-four (neuromuscular function monitor).
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Rocuronium 0.6 - 1.2 mg/kg with the dose adjusted to achieve 1-2 post-tetanic counts (Deep NMB) or 1-2 twitches in the train-on-four (Moderate NMB).
  Other Names: Zemuron

SUMMARY:
The goal of this study is to investigate the effect of depth of neuromuscular block (NMB) on global and regional (dependent versus nondependent) respiratory mechanics during laparoscopic surgery. Furthermore, we will investigate if the level of NMB influences intraoperative hemodynamic and cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Elective patients scheduled to undergo laparoscopic surgery with expected duration > 2h
* Physical status ASA I - III

Exclusion Criteria:

* Pregnancy
* Severe cardiac disease (NYHA class III or IV, acute coronary syndrome, or persistent ventricular tachyarrhythmia)
* Previous lung surgery
* History of severe chronic obstructive pulmonary disease
* Gastro-esophageal pathology (including but not limited to recent gastric or esophageal surgery including bypass/banding, history of esophageal varices, known anatomical gastric or esophageal defects such as strictures, hernias or fistulas)
* Mechanical ventilation within the last 30 days
* Neuromuscular disease
* Consented for another interventional study or refusal to participate in the present study
* Hypersensitivity (e.g., anaphylaxis) to rocuronium bromide or other neuromuscular blocking agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Vidal Melo, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Joris J, Cigarini I, Legrand M, Jacquet N, De Groote D, Franchimont P, Lamy M. Metabolic and respiratory changes after cholecystectomy performed via laparotomy or laparoscopy. Br J Anaesth. 1992 Oct;69(4):341-5. doi: 10.1093/bja/69.4.341. PMID 1419439
- [Background] Ivankovich AD, Miletich DJ, Albrecht RF, Heyman HJ, Bonnet RF. Cardiovascular effects of intraperitoneal insufflation with carbon dioxide and nitrous oxide in the dog. Anesthesiology. 1975 Mar;42(3):281-7. doi: 10.1097/00000542-197503000-00008. PMID 123134
- [Background] Dexter SP, Vucevic M, Gibson J, McMahon MJ. Hemodynamic consequences of high- and low-pressure capnoperitoneum during laparoscopic cholecystectomy. Surg Endosc. 1999 Apr;13(4):376-81. doi: 10.1007/s004649900993. PMID 10094751
- [Background] Karsten J, Heinze H, Meier T. Impact of PEEP during laparoscopic surgery on early postoperative ventilation distribution visualized by electrical impedance tomography. Minerva Anestesiol. 2014 Feb;80(2):158-66. Epub 2013 Jul 23. PMID 23877309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deep Neuromuscular Block (NMB) | Moderate Neuromuscular Block (NMB)
Started | 16 | 21
Completed | 16 | 19
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep Neuromuscular Block (NMB) | Moderate Neuromuscular Block (NMB) | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.9) | 60.7 (9.6) | 58.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 11 | 15 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 19 | 35
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (8.1) | 28.0 (4.5) | 28.3 (7.7)
ASA Physical Status Classification [Count of Participants; unit: Participants] — ASA I A normal healthy patient ASA II A patient with mild systemic disease
  Participants
    I | 1 | 2 | 3
    II | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Regional Change in Air Content (Delta Z, %)
Description: We will measure continuous respiratory flows and pressures in the intraoperative period to assess continuously the compliance and resistance of the respiratory system (T1 to T5). In addition, we will use an esophageal balloon to assess esophageal pressures and partition the global mechanical properties of the respiratory system, into their lung and chest wall components (T1 to T5). Regional lung aeration will be assessed for quantification of intraoperative lung recruitment using Electrical Impedance Tomography (EIT) (T0 to T6). Percent change was calculated using electrical impedance measurements obtained at time T0 as reference.
Time Frame: BL; During pneumoperitoneum; Stage w/2 depths neuromuscular blockade targeted - TOF1 and Deep: 1-2 twitches in post-tetanic count (50-Hz tetanus followed by three-second pause and 15 1-Hz stimuli); and immediately after release of pneumoperitoneum
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Deep Neuromuscular Block (NMB): Deep (1st) of Deep-TOF1-Deep: Deep Neuromuscular Block (NMB): Deep (1st) of Deep-TOF1-Deep group
- Deep Neuromuscular Block (NMB): MODERATE of of Deep-TOF1-Deep: Deep Neuromuscular Block (NMB): MODERATE (TOF1) of Deep-TOF1-Deep group
- Deep Neuromuscular Block (NMB): Deep (2nd) of Deep-TOF1-Deep: Deep Neuromuscular Block (NMB): Deep (2nd) of Deep-TOF1-Deep group
- Moderate Neuromuscular Block (NMB): MOD(1st) of TOF1-Deep-TOF1: Moderate Neuromuscular Block (NMB): MODERATE (1st TOF1) of TOF1-Deep-TOF1 group
- Moderate Neuromuscular Block (NMB): Deep of TOF1-Deep-TOF1: Moderate Neuromuscular Block (NMB): Deep of TOF1-Deep-TOF1 group
- Moderate Neuromuscular Block (NMB): MOD(2nd) of TOF1-Deep-TOF1: Moderate Neuromuscular Block (NMB): MODERATE (2nd TOF1) of TOF1-Deep-TOF1 group
Arm/Group | Deep Neuromuscular Block (NMB): Deep (1st) of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): MODERATE of of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): Deep (2nd) of Deep-TOF1-Deep | Moderate Neuromuscular Block (NMB): MOD(1st) of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): Deep of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): MOD(2nd) of TOF1-Deep-TOF1
Number analyzed (Participants) | 16 | 16 | 16 | 19 | 19 | 19
percent change | 14.5 (51.6) | 29.0 (43.0) | 43.3 (39.9) | -14.0 (40.2) | 19.4 (41.2) | 29.8 (38.2)

2. Primary Outcome: Ejection Fraction (%)
Description: To assess cardiac performance, transthoracic echocardiography will be used. Ejection fraction was measured as fractional shortening (FS). FS is the fraction of any diastolic dimension that is lost in systole. FS = 100*(LVEDD - LVESD) / LVEDD, LVEDD = LV end-diastolic dimension (mm); LVESD = LV end-systolic dimension (mm).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: % fractional shortening
Arm/Group | Deep Neuromuscular Block (NMB): Deep (1st) of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): MODERATE of of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): Deep (2nd) of Deep-TOF1-Deep | Moderate Neuromuscular Block (NMB): MOD(1st) of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): Deep of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): MOD(2nd) of TOF1-Deep-TOF1
Number analyzed (Participants) | 16 | 16 | 16 | 19 | 19 | 19
% fractional shortening | 36 (5) | 34 (5) | 35 (4) | 35 (5) | 36 (2) | 37 (6)

3. Primary Outcome: Cerebral Oximetry (%)
Description: Regional cerebral oxygenation will be assessed continuously during the intraoperative period using NIRS technology.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent cerebral saturation
Arm/Group | Deep Neuromuscular Block (NMB): Deep (1st) of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): MODERATE of of Deep-TOF1-Deep | Deep Neuromuscular Block (NMB): Deep (2nd) of Deep-TOF1-Deep | Moderate Neuromuscular Block (NMB): MOD(1st) of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): Deep of TOF1-Deep-TOF1 | Moderate Neuromuscular Block (NMB): MOD(2nd) of TOF1-Deep-TOF1
Number analyzed (Participants) | 16 | 16 | 16 | 19 | 19 | 19
percent cerebral saturation | 74 (6) | 73 (5) | 74 (6) | 75 (6) | 75 (6) | 75 (7)

4. Secondary Outcome: Postoperative Pain
Description: The patient will be inquired about pain with a visual analogue scale (VAS). Pain will be evaluated as incisional pain using VAS (0 = no pain; 100 = worst possible pain).
Time Frame: Postoperative Day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Deep Neuromuscular Block (NMB) | Moderate Neuromuscular Block (NMB)
Number analyzed (Participants) | 16 | 19
units on a scale | 3.5 (2.0) | 3.1 (2.2)

ADVERSE EVENTS:
Arm/Group | Deep Neuromuscular Block (NMB) | Moderate Neuromuscular Block (NMB)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes